CLINICAL TRIAL: NCT07113964
Title: QUEEN-OSCAR: A Prospective, Multicenter, Single-arm, Phase 2 Study of QL1706 in Combination With Olaparib in Previously Treated HER2-negative Breast Cancer Patients With Homologous Recombination Deficiency (HRD)
Brief Title: QL1706 With Olaparib for Previously Treated HER2-negative Breast Cancer Patients With Homologous Recombination Deficiency (HRD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-BC-IIT-002
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Previously Treated HER2-negative Breast Cancer Patients With Homologous Recombination Deficiency
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental:QL1706 + olaparib (Experimental)
  Interventions: Drug: QL1706 + olaparib

INTERVENTIONS:
Drug: QL1706 + olaparib — QL1706 is a novel dual immune checkpoint blockade containing a mixture of anti-PD1 IgG4 and anti-CTLA4 IgG1 antibodies.
  Other Names: Iparomlimab and Tuvonralimab Injection Olaparib is a poly (ADP-ribose) polymerase (PARP) inhibitor with biologic activity in ovarian cancer as well as other solid tumors..
  Other Names: NA

SUMMARY:
This study will evaluate the safety and efficacy of QL1706 and Olaparib in human epidermal growth factor receptor 2 (HER2)-negative unresectable and/or metastatic breast cancer who had received 2-4 line of prior systematic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years; Eastern Cooperative Oncology Group (ECOG) score status 0-1.
2. Pathologically documented HER2-negative locally advanced or metastatic breast cancer (IHC0, IHC 1+& IHC 2+/ISH-) that was hormone-receptor positive (i.e., estrogen-receptor positive, progesterone-receptor positive, or both) or was triple negative.
3. Has been treated with 2-4 previous therapy regimens for metastatic disease.
4. HRD positive confirmed, known germline and/or systemic BRCA mutation status that is predicted to be deleterious or suspected deleterious allow preferential enrolment.
5. At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors version 1.1.
6. Has protocol-defined adequate bone marrow, renal, hepatic and blood clotting functions.
7. A life expectancy of at least 12 weeks.
8. Female subjects of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and after the last dose for at least 3 months. Negative serum or urine pregnancy test within 7 days before study enrollment, and must be a non-lactating subject.
9. Volunteer to participate in this study and sign the informed consent.

Exclusion Criteria:

1. Has any active autoimmune disease, which may worsen when receiving immune stimulants.
2. Prior treatment with immune checkpoint inhibitors (ICI) (anti-CTLA-4, anti-PD-1, anti-PD-L1, combined therapy anti-PD-1/PD-L1 with anti-CTLA-4) or olaparib for advanced disease.
3. Has unresolved toxicities from previous anticancer therapy.
4. Has uncontrolled or significant cardiovascular disease.
5. Discontinuation of prior anti-PD-1/PD-L1/CTLA-4 therapy due to immune-related toxicity.
6. Known history or evidence of interstitial lung disease or active non-infectious pneumonitis.
7. Has received a live vaccine vaccination within 28 days before enrolment.
8. Has a known history of human immunodeficiency virus (HIV) infection.
9. Has known history of or is positive for Hepatitis B or Hepatitis C.
10. Any severe or poorly controlled systemic disease such as poorly controlled hypertension, active bleeding susceptibility or active infection, as judged by the investigator.
11. Has untreated or clinically active central nervous system metastases.
12. Female subjects who are pregnant, lactating or plan to become pregnant during the study.
13. Has any other condition that per protocol or in the opinion of the investigator is inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from the participant's first dose of study treatment to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No